CLINICAL TRIAL: NCT05991167
Title: EndeavorRx® Prospective Product Registry
Brief Title: EndeavorRx® Prospective Product Registry ("Expedition EndeavorRx")
Status: Active, not recruiting | Type: Observational
Sponsor: Akili Interactive Labs, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Akili-060
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: ADHD
Keywords: ADHD; AKL-T01; EndeavorRx; Akili; Registry
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- EndeavorRx Users: All participants with an active EndeavorRx prescription. Treatment regimen is as directed by their prescribing healthcare provider.
  Interventions: Device: EndeavorRx

INTERVENTIONS:
Device: EndeavorRx — EndeavorRx® is an FDA cleared digital therapeutic indicated to improve attention function as measured by computer-based testing in children ages 8-12 years old with primarily inattentive or combined-type attention-deficit/hyperactivity disorder (ADHD), who have a demonstrated attention issue. EndeavorRx is deployed on mobile devices and incorporates adaptive, simultaneous cognitive tasks in a consumer-grade action videogame-based platform with high-quality graphics and reward mechanisms.

SUMMARY:
The EndeavorRx Prospective Product Registry aims to collect real world data from participants receiving the digital therapeutic, EndeavorRx, under conditions of routine clinical practice.

DETAILED DESCRIPTION:
The objectives of this registry are to describe clinical and demographic characteristics, prescribing patterns, treatment patterns, and outcomes in participants treated with EndeavorRx in a real-world setting.

Patients and their caregivers will be informed about the registry as part of a series of product welcome emails following product activation. Patients/caregivers enroll into the study by providing their electronic informed consent (eConsent) and assent (eAssent). All data are captured electronically and securely through a commercial data capture platform. Participants can also invite their child's teacher to submit surveys of their observations of the child's ADHD symptoms for the study. Study activities are emailed to caregivers at baseline, 1, 2, 3, and 6-months after enrollment.

A valid and active EndeavorRx prescription is required to enroll. However, an active prescription throughout the entire 6 months of study participation is not required.

ELIGIBILITY:
Inclusion Criteria:

* Are prescribed EndeavorRx by their healthcare provider as part of routine clinical practice
* Provide informed consent/assent to participate in the registry

Exclusion Criteria:

* N/A

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients who are prescribed EndeavorRx and activates their prescription are eligible to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical and demographic characteristics | Baseline
  Socio-demographic and clinical characteristics of the registry population will be described using mean and standard deviation as well as median, minimum, maximum, and interquartile range, as appropriate for continuous variables, and counts with percentages for categorical variables. To explore changes in the profile of participants entering the registry over time, results may be stratified by enrollment date grouped by, for example, calendar month or quarter and year.
Prescribing patterns | Months 1, 2, 3, and 6
  Prescribing patterns will be summarized using count and percent of EndeavorRx prescriber types reported by registry participants. Analysis of treatment patterns will be repeated stratified by prescriber type to explore any potential differences in treatment approaches and/or adherence by prescribing healthcare provider specialty. To explore changes in prescribers over time, results may be stratified by enrollment date (e.g., calendar month or quarter and year).
Treatment patterns | Baseline, Months 1, 2, 3, and 6
  Past and current treatments for ADHD will be summarized for registry participants using counts and percentages. Adherence to EndeavorRx treatment will be assessed using gameplay data and may be defined based on number of missions and/or days played, duration of gameplay, and/or patterns of gameplay (e.g., level of effort) in relation to the values that would be expected per product instructions for use. Measures will be described using mean, standard deviation, median, minimum, maximum, and interquartile range for continuous variables, and counts with percentages for categorical variables. Adherence will be summarized overall and for time intervals after commencing treatment (e.g., weekly, monthly).
Conners 3 ADHD Index - Parent Form | Baseline, Months 1, 2, 3, and 6
  Descriptive statistics for each continuous outcome at baseline and each follow-up timepoint, as well as change from baseline at each follow-up timepoint, will be calculated. Changes in continuous outcome measures may also be assessed using linear mixed model repeated measures analyses (MMRM) to assess the effect of EndeavorRx treatment over time and adjust for potential confounding factors as necessary. Stratified analyses by treatment characteristics (e.g., concomitant ADHD medications, treatment adherence) may be conducted to examine whether changes in assessments vary with different treatment patterns.
Conners 3 ADHD Index - Teacher Form | Baseline, Months 1 and 3
  Descriptive statistics for each continuous outcome at baseline and each follow-up timepoint, as well as change from baseline at each follow-up timepoint, will be calculated. Changes in continuous outcome measures may also be assessed using linear mixed model repeated measures analyses (MMRM) to assess the effect of EndeavorRx treatment over time and adjust for potential confounding factors as necessary. Stratified analyses by treatment characteristics (e.g., concomitant ADHD medications, treatment adherence) may be conducted to examine whether changes in assessments vary with different treatment patterns.
Global Impression of Perceived Difficulties (GIPD) assessment | Baseline, Months 1, 2, 3, and 6
  Descriptive statistics for each continuous outcome at baseline and each follow-up timepoint, as well as change from baseline at each follow-up timepoint, will be calculated. Changes in continuous outcome measures may also be assessed using linear mixed model repeated measures analyses (MMRM) to assess the effect of EndeavorRx treatment over time and adjust for potential confounding factors as necessary. Stratified analyses by treatment characteristics (e.g., concomitant ADHD medications, treatment adherence) may be conducted to examine whether changes in assessments vary with different treatment patterns.
CAT-MH® ADHD module | Baseline, Months 1, 2, 3, and 6
  Descriptive statistics for each continuous outcome at baseline and each follow-up timepoint, as well as change from baseline at each follow-up timepoint, will be calculated. Changes in continuous outcome measures may also be assessed using linear mixed model repeated measures analyses (MMRM) to assess the effect of EndeavorRx treatment over time and adjust for potential confounding factors as necessary. Stratified analyses by treatment characteristics (e.g., concomitant ADHD medications, treatment adherence) may be conducted to examine whether changes in assessments vary with different treatment patterns.

CONTACTS AND LOCATIONS:
Overall Officials: Scott H Kollins, PhD, Principal Investigator — Akili Interactive Labs, Inc.
Locations (1):
- Akili Interactive Labs, Inc., Boston, Massachusetts, United States